CLINICAL TRIAL: NCT00747890
Title: The Effects of Surgical Treatment on Mild Obstructive Sleep Apnea and Its Co-morbidities
Brief Title: Surgical Treatment of Mild Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Henry Blomster, PhD, Kuopio University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: KUH5551817
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Active Comparator)
  Interventions: Procedure: Modified tonsillectomy
- II (Other)
  Interventions: Other: Lifestyle counselling by physician

INTERVENTIONS:
Procedure: Modified tonsillectomy — * Tonsillectomy
  * Uvulectomy
  * Soft palatal resection
  * Lifestyle counselling by physician: General (e.g. avoidance of smoking, alcohol drinking) and nutritional education, and sleeping positional guidance
  Arms: I
Other: Lifestyle counselling by physician — General (e.g. avoidance of smoking, alcohol drinking) and nutritional education, and sleeping positional guidance.
  Arms: II

SUMMARY:
Obstructive sleep apnea (OSA) is one of the most common sleep disorder. There are numerous conditions that are related to OSA, such as diabetes, cardiovascular diseases, and metabolic syndrome. If the patient with OSA have large tonsils, soft and largened uvula or flacid soft palate, one might benefit from operative treatment of OSA. The aim of our study is to find out whether an operative treatment is effective in mild OSA patients with carefully assessed anatomical predispositions. Our ultimate goal is to evaluate the effects of operative treatment in mild OSA itself and in the diseases related to OSA. We measure the cardiovasculary functions, symptoms, postoperative recovery, antropometry, laboratory tests, the quality of life, the quality of sleep and the inflammatory system in sleep apnea before and after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* BMI <35
* AHI 5-30 events/h
* Largened tonsils Grade ≥1

Exclusion Criteria:

* Age <18 or > 65
* BMI >35
* AHI <5 or >30
* Tonsil size < 1
* Severe nasal polyposis
* Pregnancy
* Chronic kidney, liver or thyroid disease
* Active treatment of OSA of any kind

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Apnea Hypopnea Index | One year(before and after surgery)

SECONDARY OUTCOMES:
Quality of life | One Year

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

REFERENCES:
- [Derived] Makkonen J, Blomster H, Raappana A, Markkanen S, Numminen J, Kivekas I, Valtonen O, Rautiainen M, Tuomilehto H. Adult obstructive sleep apnea treated with tonsillectomy: a randomized controlled clinical trial. Acta Otolaryngol. 2025 Oct;145(10):989-996. doi: 10.1080/00016489.2025.2557566. Epub 2025 Sep 16. PMID 40957567